CLINICAL TRIAL: NCT05700981
Title: Colon Capsule Endoscopy in Patients With Colonic Diverticulitis: a Randomized Controlled Trial
Brief Title: Colon Capsule Endoscopy in Patients With Colonic Diverticulitis
Acronym: CACODI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Odense University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CACODI trial
Record Dates: First submitted 2023-01-17; First posted 2023-01-26 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-01

CONDITIONS: Diverticulitis, Colonic
Keywords: colonic diverticulitis; capsule endoscopy; colonoscopy
MeSH Terms: conditions — Diverticulitis, Colonic | interventions — Endoscopy

STUDY DESIGN:
Intervention Model Description: A randomized controlled trials
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Colon capsule endoscopy (Experimental): Patients randomized to colon capsule endoscopy
  Interventions: Diagnostic Test: colon capsule endoscopy
- Colonoscopy (No Intervention): Patients randomized to colonoscopy

INTERVENTIONS:
Diagnostic Test: colon capsule endoscopy — Patient allocated for the intervention arm will have a CCE using the PillCam Colon 2 (Medtronic, Minneapolis, Minnesota, USA). Upon inclusion and allocation to the intervention arm patients are contacted by a dedicated CCE nurse. The course of the CCE procedure and preparations are explained thoroughly. In case of additional questions patients can contact the nurses by telephone during office hours (Monday-Friday, 8am-3pm). Before the CCE participants will have to undergo a bowel preparation procedure. The bowel preparation kit will be distributed by mail and is to be completed at home, beginning 72 hours before the CCE. The kit contains polyethylene glycol (PEG) sachets (Movicol, Norgine Danmark A/S, Herlev, Denmark), PEG solutions (MoviPrep, Norgine Danmark A/S, Herlev Denmark) and instructions on how to properly perform the preparation procedures.
  Arms: Colon capsule endoscopy

SUMMARY:
Introduction: Follow-up after colonic diverticulitis is a common indication for colonoscopy, even though studies have shown a low risk of positive findings in this population. The objective is to investigate colon capsule endoscopy (CCE) as a follow-up examination in patients with colonic diverticulitis compared to colonoscopy, on patient satisfaction and clinical performance.

Methods and Analysis: The investigators will conduct a single centre prospective randomized controlled trial. Patients seen at Odense University Hospital with acute diverticulitis confirmed by CT will be included and randomized to either follow-up by colonoscopy or CCE. Detection of suspected cancer, more than two polyps or any number of polyps larger than 9mm in CCE will generate an invitation to a diagnostic colonoscopy for biopsies or polyp removal. The investigators will compare colonoscopy and CCE regarding patient satisfaction and tolerance, the number of complete examinations, the number of patients referred to a subsequent colonoscopy after CCE and the prevalence of diverticula, polyps, cancers and other abnormal findings.

DETAILED DESCRIPTION:
Colon diverticulosis (CD) is extremely common and the prevalence seems to increase globally. The prevalence of CD increases with age and two-thirds of the adult population eventually develop CD. In the US the prevalence of CD was 32.6 % in patients aged 50-59 years and 71.4% in patients > 80 years of age. CD is often detected incidentally during optical colonoscopy (OC) or by computer tomography (CT). In approximately 25 % of patients with CD symptomatic colon diverticular disease develop typically comprising bloating, abdominal pain and change in bowel habits. Progression to diverticulitis is estimated to appear in approximately 1%. Most patients present with uncomplicated diverticulitis and are managed by general practitioners (GP) with the use of painkillers and oral antibiotics. Complicated diverticulitis due to perforation can be classified according to Hinchey et al. as a guidance to surgeon as to how conservative they can be. Hinchey level 1-2 can be managed conservatively. In the case of Hinchey level 3 and 4 it requires a laparoscopy with peritoneal lavage or laparotomy with colon resection and stoma formation, respectively. In patients presenting at the GP with intractable pain or signs of sepsis admission to hospital services is mandatory. Upon hospitalization, CT is the preferred diagnostic imaging modality in patients presenting with abdominal pain and suspected diverticulitis. If colonic diverticulitis is described as the symptoms-eliciting pathology without complications comprising abscess or bowel perforation patients are typically discharged from hospital with painkillers and offered an OC within 4-6 weeks, when the inflammation has resolved, to confirm the diverticulitis diagnosis. Routine OC after an episode of diverticulitis is recommended by the majority of international guidelines including Danish guidelines on handling of patients with diverticulitis. Due to a very low risk of malignancy in patients with diverticulitis the relevance of routine OC has been questioned in a recent review. The research in Colon Capsule Endoscopy (CCE) has evolved substantially since the introduction in 2006. More studies have reported a diagnostic yield equal to OC also in regard to larger polyps > 9 mm. In contrast to OC, CCE does not offer the possibility of biopsy or removal polyp. Hence, the ideal population for CCE needs to have low risk of findings with the need of endoscopic intervention. CCE is without pain and the risk of complications is extremely low compared to colonoscopy for which the estimated risk of major bleeding or perforation is 12 per 10,000 patients.

The investigators aimed to evaluate the effect of introducing CCE on patient satisfaction and discomfort compared to colonoscopy as a follow-up examination in patients with diverticulitis and the impact of introducing CCE on the need for subsequent colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patients above the age of 18 with in-hospital CT-diagnosed diverticulitis

Exclusion Criteria:

1. Recent imaging of the colonic mucosa and therefore no indication for renewed endoscopy, evaluated by the attending physician.
2. Colonic CT findings that require biopsy (suspected cancer) or polyp removal.
3. CT-verified stenosis in the gastrointestinal (GI) tract.
4. Cardiac pacemaker
5. Renal insufficiency
6. Pregnancy/breastfeeding
7. Allergies towards active substances administered in the trial
8. Unable to provide oral and written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Patient discomfort and preference | 6 months
  These patient-reported outcomes as well as an evaluation on patient preferences will be investigated using questionnaires

SECONDARY OUTCOMES:
Re-investigation rate | 6 months
  The number of patients randomized to colon capsule endoscopy that need to undergo a subsequent colonoscopy due to neoplastic findings or incomplete examination
Number of neoplastic lesions | 6 months
  Neoplastic lesions detected by colon capsule endoscopy or colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Bjørsum-Meyer, M.D., PhD, Principal Investigator — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Funen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Relevant anonymized data are available upon reasonable request.
  Data requesters should do the following to obtain data:
  Email the corresponding author for the paper to request the relevant data.
Supporting Information: Study Protocol
Time Frame: 1/1-2023 - 31/12-2023
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan and execution of a Data Sharing Agreement.

REFERENCES:
- [Derived] Schelde-Olesen B, Kaalby L, Deding U, Thygesen MMI, Andersen PV, Koulaouzidis A, Baatrup G, Bjorsum-Meyer T. Colon CApsule endoscopy compared to conventional COlonoscopy in patients with colonic DIverticulitis: the study protocol for a randomised controlled superiority trial (CACODI trial). BMJ Open. 2023 Oct 6;13(10):e073575. doi: 10.1136/bmjopen-2023-073575. PMID 37802611